CLINICAL TRIAL: NCT06205550
Title: Optimal Drug Therapy for the Suppression of Ventricular Arrhythmias in Andersen-Tawil Syndrome and Multifocal Ectopic Purkinje-related Premature Contractions: a Series of N-of-1 Trials
Brief Title: N-of-1 in ATS and MEPPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Christian van der Werf, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATS2023
Record Dates: First submitted 2023-12-29; First posted 2024-01-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Andersen Tawil Syndrome; Multifocal Ectopic Purkinje-related Premature Contractions
MeSH Terms: conditions — Andersen Syndrome | interventions — Flecainide; Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flecainide + beta-blocker (Active Comparator)
  Interventions: Drug: Flecainide + beta-blocker
- Flecainide monotherapy (Experimental)
  Interventions: Drug: Flecainide

INTERVENTIONS:
Drug: Flecainide — Flecainide monotherapy
  Arms: Flecainide monotherapy
Drug: Flecainide + beta-blocker — Flecainide + beta-blocker
  Arms: Flecainide + beta-blocker

SUMMARY:
Rationale: Andersen-Tawil syndrome (ATS) is a very rare heritable cardiac arrhythmia syndrome that is characterized by the triad of periodic paralysis, physical dysmorphisms, and ventricular arrhythmias, including bidirectional ventricular tachycardia (VT), polymorphic VT, and frequent multifocal premature ventricular contractions (PVCs). Multifocal ectopic Purkinje-related premature contractions (MEPPC) is a very rare syndrome characterized by frequent multifocal PVCs with relatively narrow QRS width. In both conditions, patients most often present with palpitations, but syncope and sudden cardiac arrest have also been reported. Left untreated, the large burden of PVCs can lead to PVC-induced cardiomyopathy. A number of therapeutic strategies are suggested in these conditions, but there is a lack of high-quality evidence on their efficacy.

Objective: To investigate the efficacy of various therapeutic strategies for reducing ventricular ectopy burden in patients with ATS or MEPPC.

Study design: Aggregated series of randomized, open-label N-of-1 trials. Each N-of-1 trial will consist of at least 2 treatment sets, each of which comprise two 7-day periods of treatment with therapy A and B, in a semi-randomized, counterbalanced order.

Study population: Adult patients with ATS or MEPPC on flecainide therapy.

Intervention: For ATS, flecainide monotherapy will be compared with combination therapy of flecainide and a β-blocker or calcium channel blocker. For MEPPC, flecainide monotherapy will be compared with combination therapy of flecainide and a β-blocker or calcium channel blocker (phase 1), and flecainide will be compared with quinidine (phase 2).

Main study endpoint: Ventricular ectopy burden on electrocardiographic monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following two primary diagnostic criteria A. Clinical diagnosis of ATS. Genetically confirmed diagnosis (i.e. class 4 or 5 KCNJ2 variant) is not required B. Clinical diagnosis of MEPPC and carrier of associated class 4 or 5 SCN5A variant
2. Has demonstrated a disease phenotype of ATS or MEPPC including ventricular arrhythmia burden at any point during follow-up on Holter monitor or other rhythm monitoring device (i.e. loop recorder, ECG patch)
3. Is currently treated with flecainide
4. Age ≥ 18 years

Exclusion Criteria:

* Pregnancy
* Contra-indication to study medication (see section 7.4)
* Significant structural heart disease (left ventricular ejection fraction <50%, history or signs of coronary ischemia, suspicion or definitive diagnosis of cardiomyopathy, or moderate/severe valve regurgitation)
* Suspicion or definitive diagnosis of another (heritable) arrhythmia syndrome, e.g. Brugada syndrome, early repolarization syndrome or catecholaminergic polymorphic ventricular tachycardia
* Presence of a short (<350 ms) or prolonged (>480 ms) heart-rate corrected QT interval on the resting ECG at baseline
* History of therapy refractory ventricular arrhythmia or intolerable side-effects on an adequate dose of any study medication, as determined by the treating cardiologist
* Serious known comorbid disease with a life expectancy of less than two years
* Ongoing medical condition that is deemed by the principal investigator to interfere with the conduct or assessments of the study or safety of the subjects
* Circumstances that prevent follow-up
* Inability to take orally administered tablets
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ventricular ectopy burden | 5 24-hour periods per treatment period

SECONDARY OUTCOMES:
Duration of longest ventricular tachycardia | 5 24-hour periods per treatment period

IPD SHARING:
Plan to Share IPD: No